CLINICAL TRIAL: NCT03694379
Title: Randomized Controlled Trial of Apneic Oxygenation Including Precipitous Intubations During RSI in the Emergency Department
Brief Title: Apneic Oxygenation Including Precipitous Intubations During RSI in the ED
Acronym: RAPID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not enroll enough patients
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Ilya Ostrovsky, MD, Assistant Professor of Emergency Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2018000579
Record Dates: First submitted 2018-09-11; First posted 2018-10-03 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Apneic Oxygenation; Endotracheal Intubation
Keywords: Apneic Oxygenation; Endotracheal intubation; Airway Management; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apneic Oxygenation (Experimental): Participants receiving apneic oxygenation
  Interventions: Other: Apneic oxygenation during endotracheal intubation
- No Apneic Oxygenation (No Intervention): Participants not receiving apneic oxygenation

INTERVENTIONS:
Other: Apneic oxygenation during endotracheal intubation — Providing oxygenation through nasal cannula during the apneic phase of endotracheal intubation.
  Arms: Apneic Oxygenation

SUMMARY:
This RCT is testing the efficacy of apneic oxygenation during endotracheal intubation in the emergency department. Currently the standard practice in the ED when performing endotracheal intubation is that some providers use apneic oxygenation (the application of a nasal cannula at 15LPM) throughout the intubation procedure, while others do not apply apneic oxygenation. Initial literature in the operating room showed that apneic oxygenation helps prevent desaturation during the procedure. However, the latest literature conducted in critical care settings (one study in the ICU and one in the ED) questions the efficacy of this intervention in critically ill patients; however, no harm has been shown. Our study aims to test this intervention further by adding in a special subset of patients that was excluded from prior studies, precipitous intubations, or those patients that have to be intubated quickly and cannot have adequate pre-oxygenation. We hypothesize that apneic oxygenation will be more efficacious in this subset than in the overall ED population. We will randomize patients requiring endotracheal intubation into intervention (apneic oxygenation) and control (no apneic oxygenation). We will measure the lowest arterial oxygen saturation from the start of the intubation procedure through 2 minutes after intubation is complete.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for our study will include patients 18 years or older who require emergent endotracheal intubation utilizing rapid sequence intubation (RSI) in the Emergency Department with first attempt taken by a resident or attending physician working in the emergency department. This includes Emergency Medicine attending physicians and residents as well as non-Emergency Medicine rotators (e.g.., Internal Medicine residents who are rotating through the Emergency Department).

Exclusion Criteria:

* Exclusion criteria include patients who are in cardiac arrest, or if the patient received any positive pressure ventilation (i.e, BPAP, CPAP, BVM) in the emergency department before RSI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Lowest oxygen saturation overall | Time between neuromuscular blockade and 2 minutes after completion of endotracheal intubation
  Lowest oxygen saturation between overall control and intervention groups

SECONDARY OUTCOMES:
Lowest oxygen saturation precipitous intubations | Time between neuromuscular blockade and 2 minutes after completion of endotracheal intubation
  Lowest oxygen saturation between control and intervention groups that did not receive adequate pre-oxygenation only
Lowest oxygen saturation pre-oxygenation | Time between neuromuscular blockade and 2 minutes after completion of endotracheal intubation
  Lowest oxygen saturation between control and intervention groups that did receive
Difference in baseline and final oxygen saturation | Decision to intubate through 2 minutes after completion of endotracheal intubation
Difference in oxygen saturation before and after apneic period | Initiation of neuromuscular blockade through 2 minutes after completion of endotracheal intubation
Desaturation | Initiation of neuromuscular blockade through 2 minutes after completion of endotracheal intubation
  The proportion of patients who desaturate below 90%
number of attempts | From first attempt at intubation through completion of endotracheal intubation procedure, approximately 2 minutes.
  number of times laryngoscope is placed into the mouth in an attempt to pass an endotracheal tube
Need for second operator | From first attempt at intubation through completion of endotracheal intubation procedure, approximately 2 minutes.
  A second physician had to attempt intubation
Need for additional intubating equipment | From first attempt at intubation through completion of endotracheal intubation procedure, approximately 2 minutes.
  The operator needed to change or add equipment to facilitate intubation
Esophageal intubations | From first attempt at intubation through entire ED stay, approximately 6 hours.
  The proportion of intubations that resulted in the endotracheal tube being placed in the esophagus
Procedural hypotension | Initiation of neuromuscular blockade to 2 minutes after completion of endotracheal intubation
  Proportion of became hypotensive at any point during the intubation procedure
Aspiration | Within 24 hours after intubation procedure was complete
  Proportion of patients that had evidence of aspiration
Hospital length of stay | Up to 28 days after intubation
  Number of days patient is hospitalized
Number of days intubated | Up to 28 days after intubation
In-hospital mortality | Up to 28 days after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Ostrovsky, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No